CLINICAL TRIAL: NCT01284803
Title: Feasibility and Acceptability of an Educational Intervention to Improve the Management of Depression in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2010-A00648-31; 2010/05
Record Dates: First submitted 2011-01-26; First posted 2011-01-27 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Patients With Moderate Depression,; First or Second Episode
Keywords: patients; moderate depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- experimental arm (Experimental)
  Interventions: Behavioral: an educational intervention

INTERVENTIONS:
Behavioral: an educational intervention — To elaborate an educational program for the management of depression in primary care

SUMMARY:
Qualitative study based on interviews and questionnaires with patients participating to an educational intervention to improve the management of depression in primary care.

Objective is to assess feasibility and acceptability of an educational intervention to improve the management of depression in primary care To elaborate an educational program for the management of depression in primary care.

DETAILED DESCRIPTION:
To assess feasibility and acceptability of an educational intervention to improve the management of depression in primary care To elaborate an educational program for the management of depression in primary care.

And perspectives are to elaborate an educational intervention to care depression in primary care

ELIGIBILITY:
Inclusion Criteria:

* age between 18-65y
* moderate depression (CIM 10)
* first or second episode
* able to read and understand French language

Exclusion Criteria:

* psychotic symptoms
* severe depression
* bipolar disorder
* suicide risk
* substance abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Qualitative study | 12 months
  It is a qualitative study based on interviews and questionnaires with patients participating to an educational intervention to improve the management of depression in primary care.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Lancon, Professor, Principal Investigator — APHM
Locations (1):
- Assistance Publique - Hopitaux de Marseille, Marseille, France